CLINICAL TRIAL: NCT05674370
Title: Clinical Evaluation of the GRIP Influenza and SARS-CoV-2 Point-of-care Assays Using Fresh Patient Nasal Swab Samples
Brief Title: A Study of the GRIP Influenza and SARS-CoV-2 POC Assays
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Matthew J. Binnicker, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-011258; 75A50122C00039 (Other Grant/Funding Number: United States Department of Health and Human)
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: COVID-19; Influenza
MeSH Terms: conditions — COVID-19; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Novel, graphene-based, point-of-care device (Experimental): Subjects will receive one additional nasal swab at the same time as clinical collection.
  Interventions: Device: GRIP Electronic Diagnostic Chip; Diagnostic Test: Laboratory-based nucleic acid amplification tests (NAATs)

INTERVENTIONS:
Device: GRIP Electronic Diagnostic Chip — Graphene-based point-of-care device for detection of respiratory viruses (e.g., COVID-19 and influenza) from a nasal swab
Diagnostic Test: Laboratory-based nucleic acid amplification tests (NAATs) — Polymerase Chain Reaction (PCR) analysis for detection of viruses (e.g., Roche cobas SARS-CoV-2 or influenza A/B) from nasal swab

SUMMARY:
The purpose of this research is to determine if the use of a new device can accurately detect a virus infection.

DETAILED DESCRIPTION:
GRIP has developed a novel, graphene-based detection system for potential use in point-of-care settings. This study will compare the performance of the GRIP device to routine PCR testing for detection of COVID-19 and influenza viruses. When patients present for routine testing for COVID-19 and influenza, they will also have a separate nasal swab collected that will be tested by the GRIP point-of-care device.

ELIGIBILITY:
Inclusion Criteria:

* Patients being tested for COVID 19 or Influenza

Exclusion Criteria:

* Patients < 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Binnicker, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Novel, Graphene-based, Point-of-care Device
Started | 45
Completed | 43
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Novel, Graphene-based, Point-of-care Device
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 43
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Positive Percent Agreement
Description: Percent of nasal swabs to report positive results for respiratory virus for both the GRIP device and NAAT routine clinical testing
Time Frame: One hour
Measure: Number; unit: percent of nasal swabs
Units Other Than Participants: nasal swabs
Arm/Group | Novel, Graphene-based, Point-of-care Device
Number analyzed (Participants) | 27
Number analyzed (nasal swabs) | 27
percent of nasal swabs | 52

2. Primary Outcome: Negative Percent Agreement
Description: Percent of nasal swabs to report negative results for respiratory virus for both the GRIP device and NAAT routine clinical testing
Time Frame: One hour
Measure: Number; unit: percent of nasal swabs
Units Other Than Participants: nasal swabs
Arm/Group | Novel, Graphene-based, Point-of-care Device
Number analyzed (Participants) | 27
Number analyzed (nasal swabs) | 27
percent of nasal swabs | 44

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of enrollment until completion of nasal swab, approximately one hour for each participant.
Arm/Group | Novel, Graphene-based, Point-of-care Device
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT05674370/Prot_SAP_000.pdf